CLINICAL TRIAL: NCT04387669
Title: Maneuver for Evaluating the Potential Recruitability of the Pulmonary Parenchyme in Patients With ARDS
Acronym: MERP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: 20-058
Record Dates: First submitted 2020-04-27; First posted 2020-05-14 (Actual); Last update posted 2020-05-14 (Actual); Status verified 2020-04

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: Mechanical ventilation; Recruitment maneuvers; PEEP; Respiratory mechanics; End-expiratory lung volume; Recruitability; Respiratory Distress Syndrome; Oxygenation; PaO2/FiO2 ratio; Recruitable volume; Derecruitment
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will try to define the threshold of the recruitable volume (Vrec), obtained by a derecruitment maneuver, that permit to identify patients responder or not to alveolar recruitment maneuvers.

DETAILED DESCRIPTION:
Background:

Acute respiratory distress syndrome (ARDS) is characterized by a major loss of lung volume due to alveolar flooding, atelectasis and consolidation. Alveolar recruitment maneuvers (ARM) permit to recruit non-aerated or poorly aerated lung tissue, and thus may improve gas exchange and oxygenation in patients with ARDS. However, ARM may also be harmful by overdistending the previously open lung tissue and can induce hemodynamic instability. The potential effectiveness and benefit of ARM depends on the patient's recruitability. A simple, routinely applicable bedside method to assess recruitability has been described in 2020 and is as efficient as multiple pressure-volume curves. We called it MERP for Potential for lung Recruitability Evaluation Method.

The investigators therefore propose to use this new method that determine lung recruitability as a diagnostic test to determine responder an non responder to ARM, and define a threshold.

Objectives:

The major aim is to determine the threshold of Vrec with the best sensitivity and specificity to define patient responders to alveolar recruitment maneuvers in ARDS.

The secondary objectives are :

* Evaluate the differences in morbi-mortality comparing responders and non responders to ARM
* Calculate the mean time of realization of the MERP+ARM maneuvers
* Estimate the occurence of secondary effects due to ARM (hemodynamic instability, arrhythmia, hypoxemia)

Methods:

This study will enroll at least 42 patients from the three Intensive Care Units at CHU Caen Normandy in 18 months. In all patients a MERP will be performed to determine the recruitable volume (Vrec). It consists to a brutal drop in PEEP level from 15 cmH2O to 5 cmH2O over a single breath maneuver to determine the increased end expiratory volume at the next respiratory cycle. The difference between this volume and the tidal volume represent the " measured recruitable volume " (Vmes). We can therefore calculate the predicted change in lung volume (Vcalc) by the product of respiratory system compliance at low PEEP (5 cmH20) and the change in pressure (10 cmH2O). Finally, the Vrec for each patients is the difference between the Vmes and the Vcalc.

An alveolar recruitment maneuver is then performed following the maximal alveolar recruitment method (driving pressure of 15 cmH2O, with 3 steps of PEEP 20-25-30 cmH2O) followed by a decremental PEEP procedure to determine the best PEEP. 15 minutes a posteriori, a blood gas sample permits to calculate the change in PaO2/FiO2 ratio.

Data Analysis:

The primary endpoint is to determine the threshold of Vrec that permits to identify responders to alveolar recruitment maneuvers defined by an improvement of the PaO2/FiO2 ratio > 20% 15 minutes after ARM, through ROC curve and Youden index.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe ARDS as per the Berlin definition (Partial pressure of oxygen (PaO2)/Fraction of inspired oxygen (FiO2) < 200 mmHg) and within 72h of onset, with a FiO2 > 60%
* Receiving assist/control mechanical ventilation with continuous sedation and neuromuscular blocker
* In supine position during the procedures and measurements
* Patients > 18 years of age

Exclusion Criteria:

* Patients < 18 years of age
* Pregnant woman
* Patient deprived of freedom or under a legal protective measure
* Hemodynamic instability defined as a mean arterial pressure < 65 mmHg or increasing doses of vasopressor drugs
* Pneumothorax, pneumomediastinum, pleural fistula, sub-cutaneous emphysema
* Chronic or recent severe cardiac dysfunction
* Patient with a PEEP > 15 cmH20 before inclusion
* Patient with no therapeutic perspective; candidate for palliative care exclusively or with end of life decision before inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Moderate to severe ARDS patients as per the Berlin definition
Sampling Method: Non-Probability Sample
Enrollment: 42 (Estimated)
Dates: Start 2020-04-12 (Actual); Primary Completion 2021-10-20 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Vrecruitable threshold (Vrec) | baseline
  The threshold of Vrec that permits to identify responders to alveolar recruitment maneuvers defined by an improvement of the PaO2/FiO2 ratio > 20% 15 minutes after ARM, through ROC curve and Youden index.

SECONDARY OUTCOMES:
Evaluate the differences between responders and non responders to ARM concerning the following endpoints : | 28 days
  * 28 days survival
  * ICU survival
Evaluate the differences between responders and non responders to ARM concerning the following endpoints : | 28 days
  * Free-days ventilation from day 1 to day 28
  * Number of days with moderate to severe ARDS criteria of Berlin definition
  * Length of ICU stay (Number of days)
  * Length of hospital stay (Number of days)
  * Number of days with neuromuscular blockers treatment
Calculate the mean time of realization of the MERP+ARM maneuvers | 15-20 minutes
Number of patients presenting adverse events of ARM : | 15-20 minutes
  * Cardiopulmonary arrest or arrhythmia per-ARM : acute atrial fibrillation or flutter, ventricular tachycardia, Heart rate > 150 bpm or < 60 bpm
  * Pneumothorax due to ARM
  * Hemodynamic instability (mean blood pressure < 65mmHg or systolic blood pressure < 90mmHg) during> 30s, or the need to introduce or increase vasopressor drug
  * Decrease of pulse oximetry (SpO2) < 85% for > 30 seconds

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire - CHU Caen, Caen, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen L, Brochard L. Lung volume assessment in acute respiratory distress syndrome. Curr Opin Crit Care. 2015 Jun;21(3):259-64. doi: 10.1097/MCC.0000000000000193. PMID 25827584
- [Background] Hess DR. Recruitment Maneuvers and PEEP Titration. Respir Care. 2015 Nov;60(11):1688-704. doi: 10.4187/respcare.04409. PMID 26493593
- [Background] Writing Group for the Alveolar Recruitment for Acute Respiratory Distress Syndrome Trial (ART) Investigators; Cavalcanti AB, Suzumura EA, Laranjeira LN, Paisani DM, Damiani LP, Guimaraes HP, Romano ER, Regenga MM, Taniguchi LNT, Teixeira C, Pinheiro de Oliveira R, Machado FR, Diaz-Quijano FA, Filho MSA, Maia IS, Caser EB, Filho WO, Borges MC, Martins PA, Matsui M, Ospina-Tascon GA, Giancursi TS, Giraldo-Ramirez ND, Vieira SRR, Assef MDGPL, Hasan MS, Szczeklik W, Rios F, Amato MBP, Berwanger O, Ribeiro de Carvalho CR. Effect of Lung Recruitment and Titrated Positive End-Expiratory Pressure (PEEP) vs Low PEEP on Mortality in Patients With Acute Respiratory Distress Syndrome: A Randomized Clinical Trial. JAMA. 2017 Oct 10;318(14):1335-1345. doi: 10.1001/jama.2017.14171. PMID 28973363
- [Background] Chen L, Chen GQ, Shore K, Shklar O, Martins C, Devenyi B, Lindsay P, McPhail H, Lanys A, Soliman I, Tuma M, Kim M, Porretta K, Greco P, Every H, Hayes C, Baker A, Friedrich JO, Brochard L. Implementing a bedside assessment of respiratory mechanics in patients with acute respiratory distress syndrome. Crit Care. 2017 Apr 4;21(1):84. doi: 10.1186/s13054-017-1671-8. PMID 28372575
- [Background] Chen L, Del Sorbo L, Grieco DL, Junhasavasdikul D, Rittayamai N, Soliman I, Sklar MC, Rauseo M, Ferguson ND, Fan E, Richard JM, Brochard L. Potential for Lung Recruitment Estimated by the Recruitment-to-Inflation Ratio in Acute Respiratory Distress Syndrome. A Clinical Trial. Am J Respir Crit Care Med. 2020 Jan 15;201(2):178-187. doi: 10.1164/rccm.201902-0334OC. PMID 31577153